CLINICAL TRIAL: NCT01696097
Title: The Effects of Pork vs. Chicken/Fish in a DASH Diet on Blood Pressure Regulation in Middle Aged and Older Adults (S31)
Brief Title: The Effects of Pork vs. Chicken/Fish in a DASH Diet on Blood Pressure Regulation in Middle Aged and Older Adults
Acronym: S31
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Prof. Foods and Nutrition, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1112011665; S31 Campbell Lab (Other: Purdue University)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary Counseling (Other): Pork vs. Chicken/Fish in a DASH Diet on Blood Pressure
  Interventions: Behavioral: DASH diet counseling

INTERVENTIONS:
Behavioral: DASH diet counseling — Comparison of protein source (chicken and fish vs. pork) as part of DASH diet on blood pressure regulation and blood lipids.

SUMMARY:
The purpose of this study is to determine if the source of dietary protein (pork or chicken/fish) as a part of the DASH diet affects blood pressure control in adults with high blood pressure.

DETAILED DESCRIPTION:
High blood pressure is a major risk factor for heart disease and stroke and affects 50 million people in the United States. Making healthy food choices, such as those in the DASH (Dietary Approaches to Stop Hypertension) Diet, has been shown to improve blood pressure control in people with high blood pressure. The purpose of this study is to determine if the source of dietary protein (pork or chicken/fish) as a part of the DASH diet affects blood pressure control in adults with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 40-75
* BMI 25-40 kg/m2
* systolic blood pressure 120-160 mm Hg
* diastolic blood pressure <100 mm Hg
* non-diabetic, no acute illness
* not following vigorous exercise program
* urinary continence

Exclusion Criteria:

* age <40 or >75
* BMI <25 or >40 kg/m2
* systolic blood pressure <120 or >160 mm Hg
* diastolic blood pressure >100 mm Hg
* diabetic, acute illness
* following vigorous exercise program
* urinary incontinence
* current smoker

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | After 6 weeks of following DASH diet

SECONDARY OUTCOMES:
Change in blood lipids | After 6 weeks of following DASH diet

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph. D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Sayer RD, Wright AJ, Chen N, Campbell WW. Dietary Approaches to Stop Hypertension diet retains effectiveness to reduce blood pressure when lean pork is substituted for chicken and fish as the predominant source of protein. Am J Clin Nutr. 2015 Aug;102(2):302-8. doi: 10.3945/ajcn.115.111757. Epub 2015 Jun 10. PMID 26063693
- See also: DASH eating plan info — http://dashdiet.org/